CLINICAL TRIAL: NCT03990688
Title: A Phase I, Randomised, Double-blind, Placebo-controlled Study to Assess the Effect of Multiple Oral Doses of AK3280 on Renal Function in Healthy Subjects
Brief Title: A Study to Assess the Effect of AK3280 on Renal Function in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Ark Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AK3280-4001
Record Dates: First submitted 2019-06-12; First posted 2019-06-19 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- AK3280 (Cohort 1) (Experimental): Subjects in Cohort 1 are administered with an oral dose of 100 mg AK3280 b.i.d from Day 1 to Day 14.
  Interventions: Drug: AK3280
- AK3280 (Cohort 2) (Experimental): Subjects in Cohort 2 are orally administered with AK3280 q.d. or b.i.d from Day 1 to Day 14. The dose adjustment for Cohort 2 will be based on the emerging data from previous cohort.
  Interventions: Drug: AK3280
- AK3280 (Cohort 3) (Experimental): Subjects in Cohort 3 are orally administered with AK3280 q.d. or b.i.d from Day 1 to Day 14. The dose adjustment for Cohort 3 will be based on the emerging data from previous cohorts.
  Interventions: Drug: AK3280
- Placebo (Placebo Comparator): For assessment of the Adverse Event (AE) profile, there are placebo controls in each dose cohort.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AK3280 — Active Substance: AK3280, Pharmaceutical Form: Tablet, Route of Administration: Oral
  Arms: AK3280 (Cohort 1); AK3280 (Cohort 2); AK3280 (Cohort 3)
Drug: Placebo — Active Substance: Placebo, Pharmaceutical Form: Tablet, Route of Administration: Oral
  Arms: Placebo

SUMMARY:
AK3280 is being developed to further improve the long-term efficacy and tolerability of treatment options for patients with fibrotic disorders.This study will evaluate the effect of AK3280 treatment on renal function and safety, and the PK of AK3280 compared with placebo in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give full written informed consent for participation in the study.
* Healthy male or female subject aged 18-45 years inclusive.
* Body Mass Index (BMI) ≥ 18.0 and ≤ 30.0 kg/m2。
* Clinically normal medical history, physical findings, vital signs, ECG and laboratory values at the time of screening, as judged by the Investigator in agreement with the Medical Monitor.
* With normal renal function defined as mean plasma eGFR ≥80 mL/min/1.73 m2 at screening.
* Male subjects and applicable female subjects must agree to use effective contraceptive methods to prevent drug exposure of a partner and pregnancy.

Exclusion Criteria:

* History of allergy to iohexol or other contrast media, to iodine or to shellfish.
* History of any clinically significant disease or disorder or any other condition that in the opinion of the Investigator renders them unsuitable to participate in the study.
* Regular use of any prescribed or non-prescribed medication within two weeks prior to the (first) administration of IMP.
* Any significant elevation at screening or on Day -2 of liver or urinary or serum or plasma renal test results.
* Subjects with poor venous access.
* Subjects who have smoked cigarettes (including vapour cigarettes), cigars, and/or used nicotine-containing products within 3 months prior to their screening visit.
* Positive screen for a drug of abuse or alcohol at screening or prior to administration of the IMP.
* Subjects who have not abstained from caffeine-containing beverages or products from at least 48 hours prior to screening.
* An abnormal diet within the 30 days prior to the first study drug dose.
* Any use of protein powders, xanthine and/or taurine containing energy drinks within 48 hours prior to screening.
* Blood donation (or corresponding blood loss) during the three months prior to screening.
* Employees of the study unit or their family members, students who are working in the study unit, or family members of the Investigator or Sponsor.
* Investigator considers the subject unlikely to comply with study procedures, restrictions and requirements.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2019-10-03 (Actual); Primary Completion 2020-09-09 (Actual); Study Completion 2020-09-21 (Actual)

PRIMARY OUTCOMES:
Directly measured absolute glomerular filtration rate (mGFR) results. | Days -1, 7, and 14.
  The effect of AK3280 treatment on GFR is measured by iohexol plasma clearance.
Change from baseline mGFR results. | Days 7 and 14.
  To compare the difference of effect of AK3280 treatment on GFR.

SECONDARY OUTCOMES:
Frequency, intensity, and seriousness of Adverse Events (AEs) | From Day -1 to Day 28.
  An AE can be any unfavorable and unintended sign (including an abnormal safety laboratory finding), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product.
Change in blood renal function biomarkers | Screening, Days -2, 7, 14, and 21.
  Blood renal function biomarkers include cystatin C, beta-trace protein, p-myoglobin, etc.
Change in urine renal function biomarkers | From Day -1 to Day 21.
  Urine renal function biomarkers include electrolytes, albumin, alpha1-microglobulin, etc.
Maximum Observed Plasma Concentration (Cmax) | Days 1, 7, and 14.
  The maximum observed plasma concentration of AK3280 and its major metabolite, AK3280-M2.
Concentration at the end of the dosing interval (Ctau) | Days 1, 7, and 14.
  The concentration of AK3280 and its major metabolite, AK3280-M2, at the end of the dosing interval.
trough plasma concentration (Ctrough) | Days 1, 7 and 14.
  The trough observed plasma concentration of AK3280 and its major metabolite, AK3280-M2.
trough plasma concentration (Ctrough) | Days 1, 7, and 14.
  The trough observed plasma concentration of AK3280 and its major metabolite, AK3280-M2.
Area under the plasma concentration-time curve from time zero up to time (AUC 0-t) | Days 1, 7, and 14.
  The area under the plasma concentration-time curve from time zero up to the last analytically quantifiable concentration of AK3280.

CONTACTS AND LOCATIONS:
Overall Officials: Jimmy Gu, Study Director — info@arkbiosciences.com
Locations (1):
- CTC Clinical Trial Consultants AB, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No